CLINICAL TRIAL: NCT07159230
Title: Point-of-care Multiplex PCR Test for Outpatients With Acute Respiratory Tract Infection at Risk of Severe Disease in Primary Healthcare: a Pragmatic Cluster-randomised Controlled Trial.
Brief Title: PCOT for Outpatients With Acute Respiratory Tract Infection at Risk of Severe Disease in Primary Healthcare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-KY-434
Record Dates: First submitted 2025-09-04; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Tract Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): community health care center in intervention group were provided with point-of-care multiplex PCR test (POCT) plus routine test. POCT testing was recommended for all enrolled patients presenting with acute respiratory infections who meet the predefined inclusion criteria. The therapeutic interventions were determined by health-care workers on the basis of POCT result, clinical assessment and guideline.
  Interventions: Diagnostic Test: point-of-care multiplex PCR test
- control group (No Intervention): patients in the control group will take the routine tests and receive anti-infective treatment according to clinical assessment and guideline.

INTERVENTIONS:
Diagnostic Test: point-of-care multiplex PCR test — community health care center in intervention group were provided with point-of-care multiplex PCR test (POCT) plus routine test. POCT testing was recommended for all enrolled patients presenting with acute respiratory infections who meet the predefined inclusion criteria. The therapeutic interventions were determined by health-care workers on the basis of POCT result, clinical assessment and guideline.
  Arms: intervention group

SUMMARY:
This study aims to evaluate the clinical value of point-of-care multiplex PCR testing (POCT) in guiding early diagnosis and target treatment for acute respiratory infections in primary healthcare settings.

DETAILED DESCRIPTION:
Advanced age, comorbidities, and immunosuppression are high-risk factors of severe disease in acute respiratory infections. In China, the exacerbation of population aging and increasing number of individuals with chronic comorbidities have aggravated the severity of the issue and posed a serious challenge to public health. However, insufficient pathogen diagnostic capabilities in primary healthcare prevents patients at high risk of severe disease from receiving timely and targeted treatments, potentially leading to delays in clinical management, adverse prognoses and increased economic burdens. This study aims to evaluate the clinical value of point-of-care multiplex PCR testing (POCT) in guiding early diagnosis and target treatment for acute respiratory infections in primary healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

1. Onset time<=7 days;
2. First visit;
3. Age>=18 years old;
4. Patients with acute upper respiratory tract infection with severe high-risk factors, or patients with acute lower respiratory tract infection;
5. The condition is allowed to be treated in an outpatient clinic;
6. Signed informed consent.

Exclusion Criteria:

1. The doctor judges that the disease is serious and requires hospitalization;
2. New unclear consciousness;
3. Respiratory rate>=30 beats/min;
4. Hypoxemia or respiratory failure;
5. Heart rate> 125 beats/min;
6. Systolic blood pressure < 90 or diastolic blood pressure < 60 mmHg;
7. Known active tuberculosis;
8. Pregnant and lactating women;
9. Have participated in this study within 90 days;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16868 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rates of respiratory failure and hospitalization | within 14 days after the diagnosis of acute respiratory infection

SECONDARY OUTCOMES:
Proportion of patients receiving an immediate antiviral treatment | within 1 day after the diagnosis
Proportion of patients receiving an immediate antiviral treatment by age, sex comorbidities, Immune status, season | within 1 day after the diagnosis
Proportion of patients receiving antiviral treatment | within 2 days
Proportion of patients receiving antibiotic treatment | within 2 days
Proportion of patients receiving target treatment | within 2 days
Proportion of patients receiving antibiotic treatment | within 7 days
Proportion of patients receiving target treatment | within 7 days
Proportion of patients receiving antibiotic treatment | within 14 days
Proportion of patients receiving target treatment | within 14 days
Duration of antibiotic treatment | within 14 days
Proportion of Patients Achieving Clinical Remission | within 3 days
Proportion of Patients Achieving Clinical Remission | within 7 days
Proportion of patients requiring unscheduled healthcare encounters or referrals due to clinical deterioration | within 3 days.
Proportion of patients requiring unscheduled healthcare encounters or referrals due to clinical deterioration | within 14 days
Proportion of patients requiring unscheduled healthcare encounters or referrals due to clinical deterioration | within 28 days
Proportion of patients who developed pneumonia | within 7 days
Proportion of patients who developed pneumonia | within 14 days
28-day mortality rate | within 28 days
overall cost | within 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Xincheng District Hospital, Hohhot; Genghis Khan Community Health Service Center; East Street & West Street Sub-district Community Health Service Center; East Yingxin Road Community Health Service Center and so on, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol